CLINICAL TRIAL: NCT01636518
Title: Hybrid Procedure for the Treatment of Long Standing Persistent Atrial Fibrillation - A Prospective Registry
Brief Title: Hybrid AF -- A Prospective Registry
Status: Withdrawn | Type: Observational
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Collaborators: Estech (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 13117
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial Fibrillation: Patients with Atrial Fibrillation that undergo standard of care procedure at the University of Kansas Hospital
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: Standard of Care — Standard of care procedure as determined by treating physician for Atrial Fibrillation

SUMMARY:
Atrial Fibrillation (AF) is a form of rapid irregular heart rhythm that starts in the upper chambers of the heart (called atria) and is often associated with many health problems. It can cause stroke, palpitations and heart failure. The management of long standing (chronic) AF may require additional medications and blood thinners, potentially for life. It may also require procedures where the heart is shocked with an electrical current to restore normal rhythm. Some patients require a procedure called radiofrequency ablation to address the arrhythmia.

The purpose of this registry is to collect information on patients undergoing this combination of procedures into a database, and to then use this information for scientific study to improve the treatment of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Documented effectiveness failure of at least one Vaughan-Williams Class III AAD
* Persistent AF as defined by the HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation
* Absence of significant structural heart disease as demonstrated by a transthoracic echocardiogram (TTE) of all four chambers of the heart, computed tomography (CT) scan or magnetic resonance imaging (MRI) scan within 6 months prior to enrollment
* Absence of left atrial thrombus as documented by an imaging study (e.g., TTE, transesophageal echocardiogram (TEE), thoracic CT scan, MRI, or left atrial angiography) within 30 days prior to procedure

Exclusion Criteria:

* History of longstanding persistent AF for more than 3 years
* Documented left atrial size of 60 mm or more
* Documented left ventricular ejection fraction (LVEF) less than 40%
* History of cerebrovascular disease, including stroke or transient ischemic attack (TIA) within 6 months prior to enrollment
* Significant underlying structural heart disease requiring surgical or procedural intervention within the last six months of initial procedure
* Known contraindication to anticoagulant therapy, or inability to comply with anticoagulant therapy
* Other clinical conditions precluding inclusion (e.g., organ disease, disturbances of hemostasis, etc.)
* Pregnancy, planned pregnancy (females of childbearing potential must have a negative pregnancy test prior to enrollment and agree not to become pregnant during the trial) or breastfeeding;
* Concomitant procedure planned

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing standard of care procedures to treat Atrial Fibrillation at the University of Kansas Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Outcomes of patients with persistent Atrial Fibrillation who undergo the standard of care hybrid procedure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, FACC, Principal Investigator — University of Kansas Medical Center